CLINICAL TRIAL: NCT00952614
Title: A Pilot Study of a Sustained Release Fluocinolone Implant for Treatment of Central Retinal Vein Occlusion
Brief Title: A Study of a Sustained Release Fluocinolone Implant for Treatment of Central Retinal Vein Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glenn Jaffe (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Glenn Jaffe, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007284; 7300 (Other: Duke legacy protocol ID)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Central Retinal Vein Occlusion
Keywords: retinal vein occlusion; sustained drug delivery implant; steroid; macular edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retisert for Retinal Vein Occlusion (Experimental): 0.59 mg Fluocinolone Acetonide (Retisert implant) for Retinal Vein Occlusion
  Interventions: Device: fluocinolone acetonide (Retisert Implant, Bausch and Lomb)

INTERVENTIONS:
Device: fluocinolone acetonide (Retisert Implant, Bausch and Lomb) — sustained release device consisting of 0.59 mg of fluocinolone acetonide
  Other Names: Retisert Implant, Bausch and Lomb, Rochester, NY

SUMMARY:
The purpose of this study is to determine whether a fluocinolone sustained drug delivery implant is effective in the treatment of central retinal vein occlusion that has caused persistent macular edema and decreased visual acuity.

DETAILED DESCRIPTION:
Currently there is limited treatment for macular edema and vision loss due to central retinal vein occlusion. Case reports have shown some benefit of intravitreal steroid injections in improving vision and reducing macular edema in eyes with retinal vein occlusions.

Recently, a sustained drug release steroid implant has been investigated and FDA approved to treat macular edema in patients with non-infectious uveitis, eye inflammation. This implant is placed through an incision in the eye wall and is designed to deliver a steroid, fluocinolone acetonide, for up to three years. In animal studies there was no detectable steroid seen in the blood stream.

This pilot trial will recruit individuals who have had a central retinal vein occlusion in at least one eye. If the macular edema and vision improves with an initial intravitreal injection, the eye will be considered to receive the sustained drug release device. The dosage of fluocinolone acetonide used is 0.59 mg.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to receive an implant if they met all the following criteria:

* A history of central retinal vein occlusion that had caused macular edema, based on clinical evaluation and demonstrated on fundus photography, fluorescein angiography, and optical coherence tomography (OCT)
* Macular edema at least one disc area in size that involved the fovea
* Males and non-pregnant females at least 18 years of age
* Intraocular Pressure (IOP) controlled at < 21 mmHg with no more than one topical ocular antihypertensive agent
* Ability and willingness to comply with treatment and follow up process and to understand and sign the informed consent form.
* Initially, patients with central retinal vein occlusion were not required to have previous therapy. However, the protocol was subsequently modified to require an intravitreal injection of triamcinolone acetonide > 12 weeks prior to study entry, with an initial decrease in macular edema and improvement in visual acuity and subsequent decline in visual acuity accompanied by increased macular edema. This modification was added to avoid enrolling patients who might have had a long-lasting response to a single intravitreal triamcinolone acetonide injection.

Exclusion Criteria:

* Patients are excluded if they have an allergy to fluocinolone acetonide or any component of the delivery system, a peripheral retinal detachment in the area of implantation, or media opacity precluding evaluation of study eye status.
* Patents with disciform scars of the fovea or atrophic changes of the macula that in the investigator's opinion would preclude benefit from treatment are excluded from the study.
* Female patients who were pregnant or lactating or not taking precautions to avoid pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Jaffe, MD, Principal Investigator — Duke Eye Center, DUMC
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty nine (29) participants were consented, 30 eyes. Of the 29 consented, there were 23 subjects included in the data pool of which one subject had both eyes included in the study.
Groups:
- Retisert for Retinal Vein Occlusion: 0.59 mg Fluocinolone Acetonide (Retisert implant) for Retinal Vein Occlusion
  fluocinolone acetonide (Retisert Implant, Bausch and Lomb) : sustained release device consisting of 0.59 mg of fluocinolone acetonide
Period: Overall Study
Arm/Group | Retisert for Retinal Vein Occlusion
Started | 30
Participants Started Treatment | 30 (29 subjects signed consent; 1 agreed for both eyes to enroll. 30 eyes rec'd drug delivery implant)
Completed | 23 (3 subjects died from unrelated causes, 3 were lost to follow-up & 1 had both eyes included in study.)
Not Completed | 7
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — other reason | 1

BASELINE CHARACTERISTICS:
Population: Twenty nine participants were consented. Of the 29 consented (30 eyes; one subject consented twice), 23 participants were studied and 24 eyes. Both eyes of one participant were studied
Arm/Group | Retisert for Retinal Vein Occlusion
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Acuity Using Early Treatment Diabetic Retinopathy Study (ETDRS) Charts
Description: Outcome measure based on eyes at time points with 10-letter ETDRS score improvement
Time Frame: baseline (preoperatively) to 3 years postoperatively
Measure: Mean (Full Range); unit: letters read correctly
Groups:
- Retisert for Retinal Vein Occlusion: 0.59 mg Fluocinolone Acetonide (Retisert implant) for Retinal Vein Occlusion
  fluocinolone acetonide (Retisert Implant, Bausch and Lomb) : sustained release device consisting of 0.59 mg of fluocinolone acetonide
  Measure visual acuity improvement from baseline to time periods of 1,2, and 3 years.
Arm/Group | Retisert for Retinal Vein Occlusion
Number analyzed (Participants) | 23
letters read correctly
  Change in ETDRS @ 1 year after implant | 12.5 [6 to 19]
  Change in ETDRS @ 2 years after implant | 14 [10 to 18]
  Change in ETDRS @ 3 years after implant | 13.5 [9 to 18]

2. Secondary Outcome: Improvement in Macular Edema on Optical Coherence Tomography and Color Photos
Description: Anatomic Change in reading of the size of the area of retinal thickening on color photographs and OCT. Total Macular Volume (TMV) in mm^3, is the calculated volume from the layers of the retina based off OCT imaging.
Time Frame: baseline (preoperatively) to 3 years postoperatively
Measure: Mean (Inter-Quartile Range); unit: improvement in TMV/mm^3
Arm/Group | Retisert for Retinal Vein Occlusion
Number analyzed (Participants) | 23
improvement in TMV/mm^3 | 10.4 [9.0 to 11.7]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Retisert for Retinal Vein Occlusion
Serious Adverse Events (participants affected / at risk) | 3/29
Other Adverse Events (participants affected / at risk) | 1/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Retisert for Retinal Vein Occlusion (N=29)
Death (General disorders) | 3/23 (3) — Unrelated to study activity. 29 subjects consented, 30 enrolled. 1 subject consented twice. Ocular AEs are based on 30 eyes.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retisert for Retinal Vein Occlusion (N=29)
Endophthalmitis (Infections and infestations) | 1 (1) — Developed 1 week after implant & resolved. Retinal Detachment (RD) developed months later; implant was removed during RD repair. 29 subjects consented, 30 enrolled. 1 subject consented twice. Ocular AEs are based on 30 eyes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes